CLINICAL TRIAL: NCT02278653
Title: Follow up and Functional Outcome of Organ Saving Treatment in Patients With Good Response to Neo-adjuvant (Chemo)Radiation for Rectal Cancer
Brief Title: Functional Outcome of Organ Preservation After Neo-adjuvant Chemo Radiation for Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: NL49171.068.14
Record Dates: First submitted 2014-10-06; First posted 2014-10-30 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Rectal Neoplasms
Keywords: Restaging; Watchful Waiting; Quality of Life; Manometry
MeSH Terms: conditions — Rectal Neoplasms | interventions — Surveys and Questionnaires; Manometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: The population will consist of patients, aged 18 years or older, with locally advanced rectal cancer who after chemoradiation have a clinical complete response (ycT0N0) or very good response (ycT1-2N0).
  Interventions: Other: Questionnaires for the evaluation of Quality of Life; Other: Manometry

INTERVENTIONS:
Other: Questionnaires for the evaluation of Quality of Life — 1. European Organisation for Research and Treatment of Cancer (EORTC) QLQ-30 questionnaire, version 3.0, Global Quality of Life Score
  2. Short Form (36) health survey
  3. EORTC CR38
  4. Vaizey score
  5. Low Anterior Resection Syndrome (LARS) score
  6. International Index of Erectile Function for men
  7. International Prostate Symptom Score for men
  8. Female Sexual Function Index for women
Other: Manometry — Manometry is a tool to measure the anal sphincter function. Patients do not need any bowel preparation before this procedure. During the examination a catheter tip will be positioned in the rectum above the sphincter and a small balloon will be inflated. This balloon is connected to a device that registers the measurements. Patients will receive instructions; e.g. squeeze, push, and cough. The procedure takes approximately 10 minutes and is not experienced as painful. Several parameters will be measured: the mean basal pressure, the maximum squeeze pressure, first sensation, first urge to defecate and the maximum tolerable volume. The manometric measurement will take place on the same day as the endoscopy and MRI (standard follow-up).

SUMMARY:
The primary objective is to describe the functional outcome of patients that choose for organ saving treatment.

DETAILED DESCRIPTION:
Rectal cancer is a common form of cancer. Standard treatment for locally advanced rectal cancer is a long course of neoadjuvant radiation combined with chemotherapy (CRT) followed by resection. However, neoadjuvant CRT induces downsizing and downstaging, resulting in a complete response in 15-20% of the patients. In these patients surgery may be omitted. In the investigators previous study the investigators obtained good results with an organ saving treatment. Although the mortality and morbidity associated with radical surgery is avoided, the irradiated rectum remains in situ, possibly causing functional problems.

The primary objective is to describe the functional outcome of patients that choose for organ saving treatment. Functional outcome will be evaluated with questionnaires (quality of life) and manometric measurements (maximal resting pressure, maximal squeezing pressure, sphincter length, percentage asymmetry of the resting sphincter, sustained duration, length of the high pressure zone, rectoanal inhibitory reflex, rectal sensory threshold, and rectal compliance).

Secondary objectives include: the estimation of the cumulative risk of local failure within 5 years, the estimation of the cumulative risk of disease-free, distant-metastasis-free and overall survival within 5 years, determine the percentage of patients that chooses organ saving treatment instead of standard resection, determine the compliance to intensive follow-up, and compare the cost-effectiveness of organ saving treatment to standard surgical resection over a period of 5 years. These objectives will be assessed by frequent revision of the electronic patient file, as the patient is followed up to four times per year.

Study design: prospective observational registration study with 'invasive diagnostic procedures' Study population: The population will consist of patients, aged 18 years or older, with locally advanced rectal cancer who after chemoradiation have a clinical complete response (ycT0N0) or very good response (ycT1-2N0).

Main study parameters/endpoints: The main study endpoint is the functional outcome scores based on questionnaires and manometric measurements Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The questionnaires take approximately 20 minutes to complete. There is a relatively low rate of side effects associated with manometric measurements. Results of this study will contribute to better understanding of functional complaints after rectal cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Patients with primary rectal cancer without distant metastases who underwent CRT and show clinical complete response or very good response :

  * Clinical complete response (ycT0N0) after neo-adjuvant chemoradiation will be determined clinically (digital rectal examination, endoscopy) and radiologically (contrast-enhanced-MRI)
  * Very good response (ycT1-2N0) after neo-adjuvant chemoradiation will be determined clinically (digital rectal examination, endoscopy) and radiologically (contrast-enhanced-MRI). These patients will undergo a TEM to resect the small residual tumor
* Comprehension of the alternative strategies and the concept of unknown risks are clear to the patient
* Choosing for the organ-saving treatment option (wait&see policy or TEM)
* Informed consent

Exclusion Criteria:

* Unable to understand or read Dutch
* Unwilling to comply to the questionnaires or manometric measurement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will consist of patients, aged 18 years or older, with locally advanced rectal cancer who after chemoradiation have a clinical complete response (ycT0N0) or very good response (ycT1-2N0). Patients will be recruited from the outpatient clinic, by researchers or research nurses at Maastricht University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-10 (Actual); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | 5 years
  Functional outcome scores of patients that are treated with an organ saving strategy compared to patients who undergo the standard resection as described in literature.
  Functional outcome will be evaluated with the following questionnaires:
  1. European Organisation for Research and Treatment of Cancer (EORTC) QLQ-30 questionnaire, version 3.0, Global Quality of Life Score
  2. Short Form (36) health survey
  3. EORTC CR38
  4. Vaizey score
  5. Low Anterior Resection Syndrome (LARS) score
  6. International Index of Erectile Function for men
  7. International Prostate Symptom Score for men
  8. Female Sexual Function Index for women
  Functional outcome will be measured by manometric measurements:
  1. mean basal pressure (mmH2O)
  2. maximum squeeze pressure (mmH2O)
  3. first sensation (mL)
  4. first urge to defecate (mL)
  5. maximum tolerable volume (mL)

SECONDARY OUTCOMES:
Cumulative risk of local failure | 5 years
  All patients with a local recurrence will be excluded form further follow-up. This information will be based on an MRI of the lower abdomen in combination with endoscopy.
Cumulative risks of disease-free, distant-metastasis free and overall survival | 5 years
The percentage of patients that choose the alternative strategies instead of traditional strategies and the motivation for their choice | 3 years
The compliance to the intensive follow-up schedule | 5 years
  All patients are intended to participate in the standard follow-up schedule. Some of them may drop out due to other illness, ageing or other reasons. These patients will be included in the analysis as far as they participated.
Early detection of local failure (standard surgery still possible) | 5 years
  In the first year, every three months an MRI of the lower abdomen is made in combination with an endoscopy. From the second to the fifth year, these investigations will be done twice a year. With these short intervals, it is know that local recurence is detected in an early fase.

CONTACTS AND LOCATIONS:
Overall Officials: Geerard L Beets, MD, PhD, Principal Investigator — Surgery, MUMC+; Rianne CJ Beckers, MD, MSc, Study Chair — Surgery/Radiology MUMC+; Miriam M van Heeswijk, MD, MSc, Study Chair — Surgery/Radiology MUMC+; Monique Maas, MD, PhD, Study Chair — Radiology, MUMC+
Locations (1):
- MUMC+, Maastricht, Netherlands

REFERENCES:
- [Background] Maas M, Beets-Tan RG, Lambregts DM, Lammering G, Nelemans PJ, Engelen SM, van Dam RM, Jansen RL, Sosef M, Leijtens JW, Hulsewe KW, Buijsen J, Beets GL. Wait-and-see policy for clinical complete responders after chemoradiation for rectal cancer. J Clin Oncol. 2011 Dec 10;29(35):4633-40. doi: 10.1200/JCO.2011.37.7176. Epub 2011 Nov 7. PMID 22067400
- [Background] Maas M, Nelemans PJ, Valentini V, Das P, Rodel C, Kuo LJ, Calvo FA, Garcia-Aguilar J, Glynne-Jones R, Haustermans K, Mohiuddin M, Pucciarelli S, Small W Jr, Suarez J, Theodoropoulos G, Biondo S, Beets-Tan RG, Beets GL. Long-term outcome in patients with a pathological complete response after chemoradiation for rectal cancer: a pooled analysis of individual patient data. Lancet Oncol. 2010 Sep;11(9):835-44. doi: 10.1016/S1470-2045(10)70172-8. Epub 2010 Aug 6. PMID 20692872
- [Background] Habr-Gama A, Perez RO, Proscurshim I, Campos FG, Nadalin W, Kiss D, Gama-Rodrigues J. Patterns of failure and survival for nonoperative treatment of stage c0 distal rectal cancer following neoadjuvant chemoradiation therapy. J Gastrointest Surg. 2006 Dec;10(10):1319-28; discussion 1328-9. doi: 10.1016/j.gassur.2006.09.005. PMID 17175450
- [Background] Lambregts DM, Beets GL, Maas M, Kessels AG, Bakers FC, Cappendijk VC, Engelen SM, Lahaye MJ, de Bruine AP, Lammering G, Leiner T, Verwoerd JL, Wildberger JE, Beets-Tan RG. Accuracy of gadofosveset-enhanced MRI for nodal staging and restaging in rectal cancer. Ann Surg. 2011 Mar;253(3):539-45. doi: 10.1097/SLA.0b013e31820b01f1. PMID 21239980
- [Background] Lambregts DM, Vandecaveye V, Barbaro B, Bakers FC, Lambrecht M, Maas M, Haustermans K, Valentini V, Beets GL, Beets-Tan RG. Diffusion-weighted MRI for selection of complete responders after chemoradiation for locally advanced rectal cancer: a multicenter study. Ann Surg Oncol. 2011 Aug;18(8):2224-31. doi: 10.1245/s10434-011-1607-5. Epub 2011 Feb 23. PMID 21347783
- [Background] Curvo-Semedo L, Lambregts DM, Maas M, Thywissen T, Mehsen RT, Lammering G, Beets GL, Caseiro-Alves F, Beets-Tan RG. Rectal cancer: assessment of complete response to preoperative combined radiation therapy with chemotherapy--conventional MR volumetry versus diffusion-weighted MR imaging. Radiology. 2011 Sep;260(3):734-43. doi: 10.1148/radiol.11102467. Epub 2011 Jun 14. PMID 21673229
- [Background] Habr-Gama A, Perez RO, Wynn G, Marks J, Kessler H, Gama-Rodrigues J. Complete clinical response after neoadjuvant chemoradiation therapy for distal rectal cancer: characterization of clinical and endoscopic findings for standardization. Dis Colon Rectum. 2010 Dec;53(12):1692-8. doi: 10.1007/DCR.0b013e3181f42b89. PMID 21178866
- [Background] Lambregts DM, Maas M, Bakers FC, Cappendijk VC, Lammering G, Beets GL, Beets-Tan RG. Long-term follow-up features on rectal MRI during a wait-and-see approach after a clinical complete response in patients with rectal cancer treated with chemoradiotherapy. Dis Colon Rectum. 2011 Dec;54(12):1521-8. doi: 10.1097/DCR.0b013e318232da89. PMID 22067180
- [Derived] Geubels BM, Maas M, Beets GL, Grotenhuis BA; Dutch Watch-and-Wait Consortium. What To Do With Suspected Nodal Regrowth on MRI During Follow-Up in an Organ Preservation Approach for Rectal Cancer? Dis Colon Rectum. 2024 Dec 1;67(12):1528-1535. doi: 10.1097/DCR.0000000000003385. Epub 2024 Sep 6. PMID 39250317
- [Derived] Haak HE, Zmuc J, Lambregts DMJ, Beets-Tan RGH, Melenhorst J, Beets GL, Maas M; Dutch Watch-and-Wait Consortium. The evaluation of follow-up strategies of watch-and-wait patients with a complete response after neoadjuvant therapy in rectal cancer. Colorectal Dis. 2021 Jul;23(7):1785-1792. doi: 10.1111/codi.15636. Epub 2021 Apr 2. PMID 33725387